CLINICAL TRIAL: NCT04966507
Title: A Randomized Crossover Study to Evaluate the Efficacy of Antibacterial Mouthwash in Preventing Pharyngeal Gonorrhea Among a High Risk Population
Brief Title: Antibacterial Mouthwash for Pharyngeal Gonorrhea Prevention
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Marjan Javanbakht, MPH, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: R21AI147969 (NIH); R21AI147969 (NIH)
Record Dates: First submitted 2021-05-26; First posted 2021-07-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Listerine Cool Mint Antiseptic Mouthwash (Active Comparator): Daily use of an antibacterial mouthwash (Listerine Cool Mint Antiseptic Mouthwash) during the 12-week follow-up period.
  Interventions: Drug: Listerine Antiseptic Mouthwash Product
- Biotene Oral Rinse (Placebo Comparator): Daily use of a placebo mouthwash with no known antibacterial qualities (Biotene Oral Rinse) during the 12-week follow-up period.
  Interventions: Drug: Biotene Mouthwash

INTERVENTIONS:
Drug: Listerine Antiseptic Mouthwash Product — COOL MINT LISTERINE® Antiseptic Mouthwash will be used as the 'active' study drug condition. This is a commercially available, over the counter mouthwash product. Active ingredients for this product include Eucalyptol 0.092%, Menthol 0.042%, Methyl salicylate 0.060%, Thymol 0.064%. This product also contains 21% alcohol. Participants will be asked to rinse and gargle their mouth with 20mL of mouthwash daily.
  Other Names: Active Mouthwash
  Arms: Listerine Cool Mint Antiseptic Mouthwash
Drug: Biotene Mouthwash — Biotène Rinse is designed with a moisturizing formula to help relieve dry mouth symptoms and is specifically designed to have a pH similar to saliva. This is a commercially available, over the counter mouthwash product. Biotène Mouthwash Ingredients include: Purified Water, Propylene Glycol, Hydrogenated Starch Hydrolysate, Poloxamer 407, Hydroxyethylcellulose, Sodium Benzoate, Flavor (Peppermint Oil), Benzoic Acid, Disodium Phosphate, Zinc Gluconate, Lactoferrin, Lysozyme, Lactoperoxidase, Potassium Thiocyanate, Aloe Vera Gel, Calcium Lactate, Glucose Oxidase. Participants will be asked to rinse and gargle their mouth with 20mL of mouthwash daily.
  Other Names: Placebo Mouthwash
  Arms: Biotene Oral Rinse

SUMMARY:
This study aims to determine acceptability and preliminary efficacy of daily use of an antibacterial mouthwash as compared to a placebo mouthwash in reducing the incidence of pharyngeal gonorrhea among a cohort of HIV-positive and high risk HIV-negative men.

Investigators plan to test the following hypotheses:

1. Participants will maintain a high level of adherence and satisfaction with daily mouthwash use. Furthermore, the investigators hypothesize that barriers to adherence will include structural factors such as unstable housing and individual level factors such as substance use.
2. Participants receiving the antibacterial mouthwash will have a lower incidence of pharyngeal gonorrhea as compared to participants receiving the placebo mouthwash. Furthermore, the investigators hypothesize that these reductions will remain even after adjusting for other factors such as HIV-status and substance use.

DETAILED DESCRIPTION:
The proposed study will build on the NIH/NIDA funded mSTUDY (U01 DA036267 PIs Gorbach and Shoptaw), which is a longitudinal study designed to assess the impact of substance use and HIV on minority MSM. Participants in the proposed study will be those enrolled in the mSTUDY and the objectives of this study are to measure the preliminary efficacy and acceptability of antibacterial mouthwash use for the prevention of pharyngeal gonorrhea among a cohort of high risk HIV-negative and HIV-positive MSM. In order to achieve this goal the investigators propose to conduct a double-blind, randomized, crossover trial of daily antibacterial mouthwash use as compared to a placebo mouthwash among mSTUDY participants at high risk for pharyngeal gonorrhea (i.e. previously diagnosed with pharyngeal gonorrhea). Participants will be followed for a total of 24 weeks, with each participant receiving 12-weeks of antibacterial mouthwash and 12-weeks of placebo mouthwash.

After providing written informed consent, participants will complete a computer-based questionnaire, provide biological specimen, and will be randomly allocated to their study group. The study survey will include questions that are collected as part of mSTUDY as well as questions relevant to the proposed study. Following the questionnaire, participants will provide a bio-specimen for STI testing including: (1) urine, for chlamydia and gonorrhea testing; (2) rectal and pharyngeal swabs for gonorrhea and chlamydia testing; and (3) blood, which is used for syphilis and HIV testing, and HIV-1 RNA levels (for HIV-positive).

Participants will be randomly allocated to either first receive a 12-week antibacterial mouthwash followed by 12-weeks of placebo mouthwash or start with 12-weeks of placebo mouthwash and crossover to 12-weeks of antibacterial mouthwash. The antibacterial mouthwash and placebo are commercially available products (Cool Mint Listerine® Antiseptic mouthwash and Biotene® Oral Rinse respectively) and are selected based on evidence demonstrating inhibitory effects of the antibacterial mouthwash (Cool Mint Listerine® Antiseptic mouthwash) against N. gonorrhoeae. In order to ensure concealment of study allocation and to allow for blinding, the following procedures will be instituted:

1. the investigators will generate a computerized randomization sequence (active condition first, placebo second or placebo first, active condition second). The randomization sequence will be linked to the study identification number and maintained by study staff not involved in participant contact or data management/analysis;
2. the mouthwash will be in bottles in such a way to ensure that the placebo and active product have an identical look. While the products packaging will have a similar look a label with the study ID will allow us to link the bottle to the content. At the time of study enrollment, all participants will receive a 12-week supply of mouthwash according to their randomized study group (antibacterial or placebo) and will be instructed on how to rinse and gargle with the mouthwash on a daily basis.

When participants return for the 12-week visit, they will receive another 12-week supply, which will be the crossover condition to what was assigned at baseline. Participants will be instructed to stop using any other mouthwash they may have been using prior to study enrollment. All participants will be asked to return to the study site for a 12-week follow-up visit. This visit is a study specific visit and is the only visit of the three study visits that does not overlap with an mSTUDY follow-up visit. Participants will be asked to complete a computer-based survey to collect information comparable to what was collected at baseline including information on sexual behaviors, substance use, and oral hygiene practices. Additionally, participants will be asked to complete questions regarding study mouthwash us including frequency and timing of mouthwash use (i.e., intervention fidelity) and acceptability of mouthwash. Pharyngeal swabs will be collected in order to test for gonorrhea including nucleic acid amplification testing (NAAT) and culture testing. All participants will be asked to return in 12-weeks (i.e., 24-weeks from baseline) which will coincide with an mSTUDY visit and data collection procedures from baseline will be repeated including laboratory testing for STIs and survey administration.

ELIGIBILITY:
This study will only include participants recruited as part an NIH/NIDA funded study (U01 DA036267 PIs Gorbach and Shoptaw) - the mSTUDY. By design, half of the participants are HIV-positive and half are HIV-negative and other inclusion criteria for the mSTUDY are as follows:

1. At least 18 but not older than 45 years of age on day of consent
2. Identified biologically male at birth
3. Willing to return for follow-up study visits every 6 months as long as the study is ongoing and be available to return for all study visits, barring unforeseen circumstances
4. Willing and able to provide written informed consent to take part in the study
5. Willing and able to provide adequate information for locator purposes
6. STI testing at each study visit (with reporting and treatment referral when indicated)
7. Understands and agrees to local STI reporting requirements
8. If HIV-negative at screening, report unprotected anal intercourse with a male in the past 6 months

   Additional inclusion criteria specific to this study are:
9. Currently enrolled in mSTUDY
10. mSTUDY participants who have turned 45 since enrollment in mSTUDY continue to be eligible for inclusion in this study.
11. Previously diagnosed with pharyngeal gonorrhea (while an mSTUDY participant)

Participants will be excluded from the study if:

1. Mouthwash use is contraindicated, for example because of allergies or those who may need to avoid the high alcohol content of mouthwash such as recovery alcoholics maintaining their sobriety
2. They are unwilling to stop use of their current mouthwash during the 24-week study period

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adherence and acceptability of mouthwash use | This outcome will be measured at 12-weeks post intervention.
  This outcome will be assessed using self-reported questionnaire data and will include mouthwash use in terms of number of days used, amount of mouthwash used, number of times per day, duration of gargling/rinsing; reasons for not using mouthwash, and overall experience.
Adherence and acceptability of mouthwash use | This outcome will be measured at 24-weeks post intervention.
  This outcome will be assessed using self-reported questionnaire data and will include mouthwash use in terms of number of days used, amount of mouthwash used, number of times per day, duration of gargling/rinsing; reasons for not using mouthwash, and overall experience.
Laboratory identified pharyngeal gonorrhea | This outcome will be measured at 12-weeks post intervention.
  Pharyngeal swabs will be collected for gonorrhea testing using Nucleic acid amplification testing (NAAT) with Aptima Combo 2 (GenProbe, San Diego, CA). Additionally, all participants will be asked to provide consent to access medical records in order to verify any pharyngeal gonorrhea diagnoses made during the study period but resulting from testing conducted outside of the study.
Laboratory identified pharyngeal gonorrhea | This outcome will be measured at 24-weeks post intervention.
  Pharyngeal swabs will be collected for gonorrhea testing using Nucleic acid amplification testing (NAAT) with Aptima Combo 2 (GenProbe, San Diego, CA). Additionally, all participants will be asked to provide consent to access medical records in order to verify any pharyngeal gonorrhea diagnoses made during the study period but resulting from testing conducted outside of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Javanbakht, Principal Investigator — University of California, Los Angeles
Locations (1):
- Los Angeles LGBT Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided